CLINICAL TRIAL: NCT04265625
Title: The Role of Routine Fiberoptic Bronchoscopic Guidance During Percutaneous Tracheostomy. A Prospective Randomized Trial
Brief Title: Routine Use of FIBERoptic Bronchoscopic Guidance in Percutaneous TRACHeostomy
Acronym: FIBERTRACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, José Manuel Añón, MD,PhD, Instituto de Investigación Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HULP5455
Record Dates: First submitted 2020-02-05; First posted 2020-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Complications
Keywords: Percutaneous tracheostomy; Endoscopic guidance; Fiberoptic endoscopic guidance; Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- blind tracheotomy (No Intervention): no endoscopic guidance tracheotomy
- endoscopic guidance tracheotomy (Experimental): With endoscopic guidance tracheotomy
  Interventions: Device: endoscopic guidance

INTERVENTIONS:
Device: endoscopic guidance — Percutaneous tracheotomy performed by endoscopic guidance
  Arms: endoscopic guidance tracheotomy

SUMMARY:
Tracheostomy is one of the most frequently performed techniques in intensive care units. For some authors endoscopic guide as part of the percutaneous tracheostomy (PT) might reduces the incidence of serious complications. However, for others, endoscopic guide increases the procedure cost, increases airway pressure and PaCO2 and sometimes requires the presence of another physician. International guidelines conclude that there is insufficient evidence to support the routine use of bronchoscopy during PT in order to decrease the number of complications. In addition the routine use of endoscopic guide is heterogeneous according the results of six published nation surveys. Extensive randomized trials to compare PT with endoscopic guide and without endoscopic guide are needed in order to clarify this controversial issue. This constitutes the justification of this trial.

Hypothesis: Percutaneous tracheotomy performed under endoscopic guide decreases the incidence of perioperative complications of the procedure.

DETAILED DESCRIPTION:
Background

Tracheostomy is one of the most frequently performed techniques in intensive care units (ICU). A few years after the description of the percutaneous dilatational tracheostomy (PDT), endoscopic guide as part of the technique was performed in four patients. The authors concluded that the endoscopic guide provided advantages to the realization of PDT. Other authors have state that endoscopy, significantly reduces the incidence of serious complications such as posterior tracheal tears, false passage, pneumothorax and subcutaneous emphysema. However, currently endoscopic guide as part of the percutaneous tracheostomy is controversial. Although for some authors its use reduces the number of complications, others found that endoscopic guide increases the procedure cost, increases airway pressure and PaCO2 and sometimes requires the presence of another physician. Thus, some do not consider it necessary when the physicians have enough experience with percutaneous tracheostomy. International guidelines conclude that there is insufficient evidence to support the routine use of bronchoscopy during percutaneous tracheostomy in order to decrease the number of complications. In addition the routine use of endoscopic guide is heterogeneous according the published surveys. Specifically, in Spain its use was the lowest of the six published nation surveys. Extensive randomized trials to compare percutaneous tracheostomy with endoscopic guide and without endoscopic guide are needed in order to clarify this controversial issue. This constitutes the justification of this trial.

Hypothesis

Percutaneous tracheostomy performed under endoscopic control does not reduce the incidence of perioperative complications of the procedure in critically ill patients when it is performed by experienced physicians in patients without anatomical abnormalities.

Main goal

1. - To assess the incidence of perioperative complications of percutaneous tracheotomy under endoscopic guide versus blind percutaneous tracheotomy.
2. - To assess the ventilatory parameters during percutaneous tracheostomy with and without endoscopic control.

Methodology

Prospective, multicenter randomized study. Patients admitted to the ICU who need tracheostomy due to prolonged mechanical ventilation, who do not have neither contraindications to perform the percutaneous technique nor contraindications to perform fibrobronchoscopy will be randomized.

The percutaneous tracheostomy will be carried out with the single-step dilation method. For its realization, the usual protocol will be followed.

The included patients will be randomized 1:1 (percutaneous tracheostomy with endoscopic guide vs percutaneous tracheostomy without endoscopic guide). The randomization system will be by closed envelope. A sample size of 221 patients in each branch has been calculated.

The percutaneous tracheostomy and fiberoptic bronchoscopy will be performed by staff with experience with both procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old requiring tracheotomy due to prolonged mechanical ventilation
* That Family members or legal representatives have signed the information sheet and informed consent

Exclusion Criteria:

* Patients with increased intracranial pressure according to intracranial pressure monitoring or suspected.
* Patients who have any absolute or relative contraindication for the percutaneous tracheostomy realization
* Patients with difficult airway

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2019-12-07 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with bleeding | From date of randomization until 24 hours later
  Bleeding with haemodynamic derangement or needing surgical review or transfusion of packed red cells.
Number of patients with hypoxemia | From date of randomization until 24 hours later
  Hypoxemia: Oxygen arterial saturation (SaO2) < 85% during more than 90 seconds and/or arrhythmia or cardiac arrest related to hypoxemia.
Number of patients in whom a loss of airway has ocurred | From randomization until the end of the procedure
  Loss of airway: Failure to be able to access the airway > 30 seconds.
Number of patients with atelectasis | From date of randomization until 24 hours later
  Atelectasis: Total or partial lung collapse not present before the technique, evidenced at postoperative control.
Number of patients with hypotension | From randomization until the end of the procedure
  Hypotension requiring treatment with vasopressors or >1000 ml of fluids during the procedure.
Number of patients with barotrauma | From date of randomization until 24 hours later
  Barotrauma: Subcutaneous emphysema, mediastinal emphysema or pneumothorax related to the technique.
Number of patients with posterior tracheal wall injury | From date of randomization until 24 hours later
  Posterior tracheal wall injury: Injury to membranous trachea by the needle, guide or dilator along with any related consequences (pneumomediastinum, pneumothorax, subcutaneous emphysema, tracheo-esophageal fistula)
Number of patients in whom false passage has ocurred | From randomization until the end of the procedure
  False passage: Dilatation or insertion of the cannula out of the trachea lumen.
Number of patients in whom cardiac arrest or death directly related to any complication arising from the technique occurred | From date of randomization until the ICU discharge
  Cardiac arrest or death

SECONDARY OUTCOMES:
Peak airway pressure | From randomization until the end of the procedure
  Maximum peak airway pressure (cmH2O)
Plateau pressure | From randomization until the end of the procedure
  Maximum plateau pressure (cmH2O)
Tidal volume | From randomization until the end of the procedure
  Minimum tidal volume (mL)
Arterial Blood Gas | From randomization until 15 minutes after the procedure
  Arterial blood gase at the beginning and the end of the procedure
Oxygen saturation (SaO2) | From randomization until the end of the procedure
  Minimum arterial oxygen saturation (SaO2)

OTHER OUTCOMES:
Mortality | From the date of randomization until the hospital discharge
  All-cause mortality at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jose Manuel Añon, MD. PhD, Principal Investigator — Hospital Universitario La Paz. IdiPAZ
Locations (4):
- Spain (4):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Rey Juan Carlos, Madrid
  - Hospital Universitario de Toledo, Toledo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anon JM, Arellano MS, Perez-Marquez M, Diaz-Alvarino C, Marquez-Alonso JA, Rodriguez-Pelaez J, Nanwani-Nanwani K, Martin-Pellicer A, Civantos B, Lopez-Fernandez A, Seises I, Garcia-Nerin J, Figueira JC, Casero H, Vejo J, Agrifoglio A, Cachafeiro L, Diaz-Almiron M, Villar J. The role of routine FIBERoptic bronchoscopy monitoring during percutaneous dilatational TRACHeostomy (FIBERTRACH): a study protocol for a randomized, controlled clinical trial. Trials. 2021 Jun 29;22(1):423. doi: 10.1186/s13063-021-05370-x. PMID 34187554
- See also: https://pubmed.ncbi.nlm.nih.gov/34187554/ — https://pubmed.ncbi.nlm.nih.gov/34187554/